CLINICAL TRIAL: NCT05752019
Title: TAAI Erasmus Research Initiative to Fight CF: Monitoring Inflammation in CF Lung Disease Into a New Era
Acronym: TERRIFIC-MILE
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Stichting TAAI (Other)
Responsible Party: Principal Investigator, Hettie M Janssens, MD PhD, Pediatric pulmonologist, Erasmus Medical Center
Other Study IDs: V2.1, 12-08-2022; MEC-2021-0907 (Other: Medical ethics committee)
Record Dates: First submitted 2022-11-15; First posted 2023-03-02 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2023-09

CONDITIONS: Cystic Fibrosis; Lung Inflammation; Lung Infection; Lung Disease; Cystic; Lung Diseases; Lung Disease; Cystic, Congenital; Inflammation Lungs; Congenital Disorders; Exacerbation, Symptom; Infections, Bacterial
Keywords: Breathomics; Exhaled Breath Analysis; Biomarkers; elexacaftor/tezacaftor/ivacaftor; Trikafta; Kaftrio; Non-invasive monitoring; Minimal-invasive monitoring; Sputum
MeSH Terms: conditions — Cystic Fibrosis; Pneumonia; Cystic Disease Of Lung; Lung Diseases; Cystic Adenomatoid Malformation of Lung, Congenital; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Symptom Flare Up; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For this study we are collecting sputum, blood, exhaled breath and urine. Patients can opt out for each sample, except exhaled breath. These specimens will be collected at each study visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- ETI treatment group > 12 years: CF patients older than 12, whom are eligible to receive elexacaftor/tezacaftor/ivacaftor treatment.
- Control group > 12 years: CF patients older than 12, whom are not eligible to receive any CFTR-modulator.
- ETI treatment group < 12 years: CF patients younger than 12, whom are eligible to receive elexacaftor/tezacaftor/ivacaftor treatment.
- Control group < 12 years: CF patients younger than 12, whom are not eligible to receive any CFTR-modulator.

SUMMARY:
Progressive destruction of the lungs is the main cause of shortened life expectancy in people with cystic fibrosis (pwCF). Inflammation and respiratory infections play a key role in CF lung disease. Previous studies have shown that an increase in inflammatory markers predicts structural lung damage. Close monitoring of pwCF is crucial to adequately provide optimal care. Pulmonary management for pwCF involves treating infections and exacerbations and promoting exercise and mucociliary clearance to slow or prevent structural lung damage. To evaluate the treatment and incite timely interventions it is important for the pulmonary physician to be well-informed about the condition of the lungs.

The main monitoring tools in regular CF care are lung function, sputum cultures, symptom reporting and more recently imaging by chest computed tomography (CT-scan) or magnetic resonance imaging (MRI). Strangely enough, there are currently no monitoring tools used in clinics to measure inflammation in the lung, although this is a main factor for progressive lung disease.

New highly effective modulator therapy (HEMT) such as elexacaftor/tezacaftor/ivacaftor [ETI, Kaftrio®] is transforming CF treatment, vastly improving lung function and reducing exacerbations. Initial CFTR modulators like ivacaftor and lumacaftor/ivacaftor also improved lung function and reduced exacerbations, but studies showed that lung inflammation was still present. The long-term impact of ETI and its effect on inflammation is not yet known.

Thus, monitoring pwCF on HEMT may be different from before, as lung damage seen on chest CT will be less apparent and lung function will improve considerably, therefore not being adequate markers for subtle changes in the lungs. Thus, the focus of monitoring in the era of highly effective CFTR modulators needs to change preferably focusing on measuring lung inflammation.

An ideal monitoring tool for lung inflammation in pwCF should be non-invasive, efficient, and provide accurate and sensitive results. Currently, sputum and BAL are the most common methods for assessing inflammation, but BAL is invasive and sputum may not always be available. Exhaled breath analysis by the electronic nose (eNose) or gas chromatography-mass spectrometry (GC-MS) of volatile organic compounds (VOCs) shows promise as a non-invasive monitoring tool. Other promising markers and techniques are inflammatory markers in the blood (cytokines and micro-RNA (miRNA)) and urine.

Thus, the objective of this project is to design novel, minimally invasive monitoring techniques capable of identifying lung inflammation in pwCF undergoing highly effective CFTR modulator therapy (ETI) compared to those not using CFTR modulators. The efficacy of these innovative techniques will be evaluated and verified against inflammatory markers in sputum, spirometry, and validated symptom and quality of life scores.

DETAILED DESCRIPTION:
Objective:

The overall aim of the study is to develop innovative minimally invasive monitoring techniques that can identify lung inflammation in pwCF when using highly effective modulators, compared to patients whom are not eligible for CFTR modulators (control group) yet.

Primary objective is to assess whether measuring VOCs with GC-MS is a sensitive method to monitor changes in lung inflammation in pwCF.

Secondary objectives are:

* To assess whether eNose is a sensitive method to monitor changes in lung inflammation in pwCF.
* To explore the usefulness of other inflammatory markers in blood and urine.

Study design: Explorative cohort study aimed to develop innovative minimally invasive monitoring techniques that can identify lung inflammation in pwCF when using highly effective CFTR modulators. (eNose, GC-MS, inflammatory markers in urine and blood), compared to a control group: pwCF not using CFTR modulators. Furthermore, the investigators will compare these techniques with inflammatory markers in induced sputum, conventional spirometry, symptom and quality of life scores.

Study population: pwCF older than 6 years of age who are eligible to start on ETI treatment and as a control group pwCF who are not on CFTR modulators,

Intervention: Subjects will be included till at least 3 study visits have taken place during treatment with ETI or for the control group: 3 consecutive regular outpatient clinic visits, which are usually 3 months apart. If the subject has not started with ETI an extra visit at baseline will be added just before start of ETI. At the study visits routine care checks will be done, such as spirometry and blood sampling for liver enzyme monitoring. The extra investigations performed at these study visits are: exhaled breath sampling, 3 extra vials of blood, urine collection, induced sputum. Lung clearance index (LCI) will be done for subjects below 18 years of age. Subjects may opt out for blood, induced sputum and urine samples, there always need to be an exhaled breath sampling with eNose and GC-MS. If the patient has a contra-indication or does not want to participate in the induced sputum procedure, the investigators will attempt to collect spontaneous expectorated sputum instead.

To limit their burden of the study for the age group 6-11, the investigators will not conduct all measurements in that age group. Resulting, in the following difference in study design between two age groups:

Patients >12 years: At all visits there will be exhaled breath sampling, 3 extra vials of blood with a blooddraw, induced sputum, urine sample and 2 questionnaires (QoL and symptom score).

Patients <12 years: At all visits there will be exhaled breath sampling and 1 questionnaire (symptom score) will be done by doing an interview with the child. On the last visit 2 extra vials of blood will be collected. For patients 6-18 years of age a multiple breath washout (MBW) for LCI will be scheduled at study visits.

Main study parameters/endpoints:

Primary endpoint is the comparison of VOCs, measured by GC-MS, during ETI treatment compared to control group over time during 3 different study visits.

Secondary endpoints entail the correlation of VOCs by GC-MS breath profiles/VOCs, measured by eNose, inflammatory markers in induced sputum (IL-8, free neutrophilic elastase (NE), calprotectin and myeloperoxidase, plus a predetermined cytokine panel), blood (IL-18, IL-1β, TNF, hsCRP, sCD14, calprotectin, HGMB-1, amyloid and miRNA), urine and, lung function, quality of life and symptom scores at baseline (if available) and overtime during 3 consecutive study visits. In addition, the change of VOCs by GC-MS and eNose from baseline till 3 months of ETI treatment will be investigated.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

Diagnosed with CF, either by abnormal sweat test and/or confirmed with 2 CF causing mutations found by genetic analysis, either from heel-prick screening or diagnosed later in life. Aged >6 years (i.e. children and adults). Age appropriate written informed consent is required.

In addition, patients need to meet the criteria of one of the following study groups:

Group 1: Treated group : people with CF with mutations who are eligible to start ETI or who are already using it. This maybe patients who transition from another CFTR modulator or who are CFTR modulator naïve.

Group 2: Control group: people with CF whom are not eligible to start on any CFTR modulator yet and receive standard treatment. This group will function as controls.

Exclusion Criteria:

- People with CF who cannot follow instructions

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: people with CF older than 6 years of age who are eligible to start on ETI treatment and as a control group people with CF who are not on CFTR modulators.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation of the peak intensities of Volatile Organic Compounds, measured by GC-MS and eNose, with inflammatory markers in sputum, like IL-8. | Study completion will take an average of 1 year.
  Correlation of Volatile Organic Compounds (VOCs), measured by GC-MS and eNose breath profiles/VOCs, with inflammatory markers in induced sputum (IL-8, free neutrophilic elastase (NE), calprotectin and myeloperoxidase, plus a predetermined cytokine panel). Volatile organic compounds are measured by gas chromatography - mass spectrometry (GC-MS) and eNose. With the GC-MS, Compounds in breath will be identified according to their retention time and m/z ratio. Difference between peak intensities of compounds will be assessed between groups. An untargeted analysis approach will be used to identify compounds that have the most discriminative ability between the defined groups.
  The sensors in the eNose will change their electric output when a participant breathes through the machine. The change in signal per sensor will be used to correlate with inflammatory markers in sputum and to identify clusters with higher and lower lung inflammation profile.

SECONDARY OUTCOMES:
Correlation of VOCs, measured by GC-MS and eNose, with validated questionnaires | Study completion will take an average of 1 year.
  Correlation of VOCs by GC-MS and eNose breath profiles/VOCs with validated questionnaires (CFRSD-CRISS & CFQ-R). CFRSD-CRISS is symptom score questionnaire and the CFQ-R a quality of life questionnaire. Both questionnaires result in certain scores, which will be used for the analysis and validation of the breath analyzing techniques. Volatile organic compounds are analyzed with GC-MS and eNose as described at the primary outcome.
Correlation of potential biomarkers in blood and urine with inflammatory markers in sputum, VOCs in Exhaled Breath and validated questionnaires. | Study completion will take an average of 1 year.
  The targeted biomarkers are listed in the study description.
Change in volatile organic compounds (VOCs), measured by GC-MS, during ETI treatment compared to control group over time. | Study completion will take an average of 1 year.
  Volatile organic compounds are measured by gas chromatography - mass spectrometry. Compounds in breath will be identified according to their retention time and m/z ratio. Difference between peak intensities of compounds will be assessed between groups. A untargeted analysis approach will be used to identify compounds that have the most discriminative ability between the defined groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC - Sophia Children's Hospital, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Background] De Boeck K. Cystic fibrosis in the year 2020: A disease with a new face. Acta Paediatr. 2020 May;109(5):893-899. doi: 10.1111/apa.15155. Epub 2020 Jan 22. PMID 31899933
- [Background] Horati H, Janssens HM, Margaroli C, Veltman M, Stolarczyk M, Kilgore MB, Chou J, Peng L, Tiddens HAMW, Chandler JD, Tirouvanziam R, Scholte BJ. Airway profile of bioactive lipids predicts early progression of lung disease in cystic fibrosis. J Cyst Fibros. 2020 Nov;19(6):902-909. doi: 10.1016/j.jcf.2020.01.010. Epub 2020 Feb 10. PMID 32057679
- [Background] Sly PD, Gangell CL, Chen L, Ware RS, Ranganathan S, Mott LS, Murray CP, Stick SM; AREST CF Investigators. Risk factors for bronchiectasis in children with cystic fibrosis. N Engl J Med. 2013 May 23;368(21):1963-70. doi: 10.1056/NEJMoa1301725. PMID 23692169
- [Background] Wijker NE, Vidmar S, Grimwood K, Sly PD, Byrnes CA, Carlin JB, Cooper PJ, Robertson CF, Massie RJ, Kemner van de Corput MPC, Cheney J, Tiddens HAWM, Wainwright CE; Australasian Cystic Fibrosis Bronchoalveolar Lavage (ACFBAL) and Follow-up of the ACFBAL (CF-FAB) study groups; following investigators constitute the ACFBAL Study Investigators Group:; following investigators constitute the CF FAB Study Investigators Group:; Additional contributions: We are indebted to all current and former clinical and research staff from Queensland Children's Hospital, Brisbane:. Early markers of cystic fibrosis structural lung disease: follow-up of the ACFBAL cohort. Eur Respir J. 2020 Apr 3;55(4):1901694. doi: 10.1183/13993003.01694-2019. Print 2020 Apr. PMID 31949117
- [Background] Smyth AR, Bell SC, Bojcin S, Bryon M, Duff A, Flume P, Kashirskaya N, Munck A, Ratjen F, Schwarzenberg SJ, Sermet-Gaudelus I, Southern KW, Taccetti G, Ullrich G, Wolfe S; European Cystic Fibrosis Society. European Cystic Fibrosis Society Standards of Care: Best Practice guidelines. J Cyst Fibros. 2014 May;13 Suppl 1:S23-42. doi: 10.1016/j.jcf.2014.03.010. PMID 24856775
- [Background] Margaroli C, Garratt LW, Horati H, Dittrich AS, Rosenow T, Montgomery ST, Frey DL, Brown MR, Schultz C, Guglani L, Kicic A, Peng L, Scholte BJ, Mall MA, Janssens HM, Stick SM, Tirouvanziam R. Elastase Exocytosis by Airway Neutrophils Is Associated with Early Lung Damage in Children with Cystic Fibrosis. Am J Respir Crit Care Med. 2019 Apr 1;199(7):873-881. doi: 10.1164/rccm.201803-0442OC. PMID 30281324
- [Background] Heijerman HGM, McKone EF, Downey DG, Van Braeckel E, Rowe SM, Tullis E, Mall MA, Welter JJ, Ramsey BW, McKee CM, Marigowda G, Moskowitz SM, Waltz D, Sosnay PR, Simard C, Ahluwalia N, Xuan F, Zhang Y, Taylor-Cousar JL, McCoy KS; VX17-445-103 Trial Group. Efficacy and safety of the elexacaftor plus tezacaftor plus ivacaftor combination regimen in people with cystic fibrosis homozygous for the F508del mutation: a double-blind, randomised, phase 3 trial. Lancet. 2019 Nov 23;394(10212):1940-1948. doi: 10.1016/S0140-6736(19)32597-8. Epub 2019 Oct 31. PMID 31679946
- [Background] Middleton PG, Mall MA, Drevinek P, Lands LC, McKone EF, Polineni D, Ramsey BW, Taylor-Cousar JL, Tullis E, Vermeulen F, Marigowda G, McKee CM, Moskowitz SM, Nair N, Savage J, Simard C, Tian S, Waltz D, Xuan F, Rowe SM, Jain R; VX17-445-102 Study Group. Elexacaftor-Tezacaftor-Ivacaftor for Cystic Fibrosis with a Single Phe508del Allele. N Engl J Med. 2019 Nov 7;381(19):1809-1819. doi: 10.1056/NEJMoa1908639. Epub 2019 Oct 31. PMID 31697873
- [Background] Jarosz-Griffiths HH, Scambler T, Wong CH, Lara-Reyna S, Holbrook J, Martinon F, Savic S, Whitaker P, Etherington C, Spoletini G, Clifton I, Mehta A, McDermott MF, Peckham D. Different CFTR modulator combinations downregulate inflammation differently in cystic fibrosis. Elife. 2020 Mar 2;9:e54556. doi: 10.7554/eLife.54556. PMID 32118580
- [Background] Fens N, van der Schee MP, Brinkman P, Sterk PJ. Exhaled breath analysis by electronic nose in airways disease. Established issues and key questions. Clin Exp Allergy. 2013 Jul;43(7):705-15. doi: 10.1111/cea.12052. PMID 23786277
- [Background] de Vries R, Dagelet YWF, Spoor P, Snoey E, Jak PMC, Brinkman P, Dijkers E, Bootsma SK, Elskamp F, de Jongh FHC, Haarman EG, In 't Veen JCCM, Maitland-van der Zee AH, Sterk PJ. Clinical and inflammatory phenotyping by breathomics in chronic airway diseases irrespective of the diagnostic label. Eur Respir J. 2018 Jan 11;51(1):1701817. doi: 10.1183/13993003.01817-2017. Print 2018 Jan. PMID 29326334
- [Background] Sagel SD, Kapsner RK, Osberg I. Induced sputum matrix metalloproteinase-9 correlates with lung function and airway inflammation in children with cystic fibrosis. Pediatr Pulmonol. 2005 Mar;39(3):224-32. doi: 10.1002/ppul.20165. PMID 15635615
- [Background] Thomassen JC, Trojan T, Walz M, Vohlen C, Fink G, Rietschel E, Alejandre Alcazar MA, van Koningsbruggen-Rietschel S. Reduced neutrophil elastase inhibitor elafin and elevated transforming growth factor-beta1 are linked to inflammatory response in sputum of cystic fibrosis patients with Pseudomonas aeruginosa. ERJ Open Res. 2021 Jul 19;7(3):00636-2020. doi: 10.1183/23120541.00636-2020. eCollection 2021 Jul. PMID 34291109
- [Background] Jain R, Baines A, Khan U, Wagner BD, Sagel SD. Evaluation of airway and circulating inflammatory biomarkers for cystic fibrosis drug development. J Cyst Fibros. 2021 Jan;20(1):50-56. doi: 10.1016/j.jcf.2020.06.017. Epub 2020 Jul 1. PMID 32622665
- [Background] Quon BS, Ngan DA, Wilcox PG, Man SF, Sin DD. Plasma sCD14 as a biomarker to predict pulmonary exacerbations in cystic fibrosis. PLoS One. 2014 Feb 20;9(2):e89341. doi: 10.1371/journal.pone.0089341. eCollection 2014. PMID 24586701
- [Background] Stachowiak Z, Wojsyk-Banaszak I, Jonczyk-Potoczna K, Narozna B, Langwinski W, Kycler Z, Sobkowiak P, Breborowicz A, Szczepankiewicz A. MiRNA Expression Profile in the Airways is Altered during Pulmonary Exacerbation in Children with Cystic Fibrosis-A Preliminary Report. J Clin Med. 2020 Jun 16;9(6):1887. doi: 10.3390/jcm9061887. PMID 32560275
- [Background] Bhattacharyya S, Balakathiresan NS, Dalgard C, Gutti U, Armistead D, Jozwik C, Srivastava M, Pollard HB, Biswas R. Elevated miR-155 promotes inflammation in cystic fibrosis by driving hyperexpression of interleukin-8. J Biol Chem. 2011 Apr 1;286(13):11604-15. doi: 10.1074/jbc.M110.198390. Epub 2011 Jan 31. PMID 21282106
- [Background] Krause K, Kopp BT, Tazi MF, Caution K, Hamilton K, Badr A, Shrestha C, Tumin D, Hayes D Jr, Robledo-Avila F, Hall-Stoodley L, Klamer BG, Zhang X, Partida-Sanchez S, Parinandi NL, Kirkby SE, Dakhlallah D, McCoy KS, Cormet-Boyaka E, Amer AO. The expression of Mirc1/Mir17-92 cluster in sputum samples correlates with pulmonary exacerbations in cystic fibrosis patients. J Cyst Fibros. 2018 Jul;17(4):454-461. doi: 10.1016/j.jcf.2017.11.005. Epub 2017 Dec 11. PMID 29241629
- [Background] Laguna TA, Wagner BD, Starcher B, Luckey Tarro HK, Mann SA, Sagel SD, Accurso FJ. Urinary desmosine: a biomarker of structural lung injury during CF pulmonary exacerbation. Pediatr Pulmonol. 2012 Sep;47(9):856-63. doi: 10.1002/ppul.22525. Epub 2012 Mar 19. PMID 22431382
- [Background] Bruce MC, Poncz L, Klinger JD, Stern RC, Tomashefski JF Jr, Dearborn DG. Biochemical and pathologic evidence for proteolytic destruction of lung connective tissue in cystic fibrosis. Am Rev Respir Dis. 1985 Sep;132(3):529-35. doi: 10.1164/arrd.1985.132.3.529. PMID 3898942
- [Background] Sampson AP, Spencer DA, Green CP, Piper PJ, Price JF. Leukotrienes in the sputum and urine of cystic fibrosis children. Br J Clin Pharmacol. 1990 Dec;30(6):861-9. doi: 10.1111/j.1365-2125.1990.tb05452.x. PMID 1963072
- [Background] Laguna TA, Williams CB, Nunez MG, Welchlin-Bradford C, Moen CE, Reilly CS, Wendt CH. Biomarkers of inflammation in infants with cystic fibrosis. Respir Res. 2018 Jan 8;19(1):6. doi: 10.1186/s12931-017-0713-8. PMID 29310632
- [Background] Martin SL, Moffitt KL, McDowell A, Greenan C, Bright-Thomas RJ, Jones AM, Webb AK, Elborn JS. Association of airway cathepsin B and S with inflammation in cystic fibrosis. Pediatr Pulmonol. 2010 Sep;45(9):860-8. doi: 10.1002/ppul.21274. PMID 20632407
- [Background] Neerincx AH, Whiteson K, Phan JL, Brinkman P, Abdel-Aziz MI, Weersink EJM, Altenburg J, Majoor CJ, Maitland-van der Zee AH, Bos LDJ. Lumacaftor/ivacaftor changes the lung microbiome and metabolome in cystic fibrosis patients. ERJ Open Res. 2021 Apr 19;7(2):00731-2020. doi: 10.1183/23120541.00731-2020. eCollection 2021 Apr. PMID 33898610
- [Background] Quittner AL, Modi AC, Wainwright C, Otto K, Kirihara J, Montgomery AB. Determination of the minimal clinically important difference scores for the Cystic Fibrosis Questionnaire-Revised respiratory symptom scale in two populations of patients with cystic fibrosis and chronic Pseudomonas aeruginosa airway infection. Chest. 2009 Jun;135(6):1610-1618. doi: 10.1378/chest.08-1190. Epub 2009 May 15. PMID 19447923
- [Background] Gold LS, Patrick DL, Hansen RN, Goss CH, Kessler L. Correspondence between lung function and symptom measures from the Cystic Fibrosis Respiratory Symptom Diary-Chronic Respiratory Infection Symptom Score (CFRSD-CRISS). J Cyst Fibros. 2019 Nov;18(6):886-893. doi: 10.1016/j.jcf.2019.05.009. Epub 2019 May 22. PMID 31126901